CLINICAL TRIAL: NCT00618917
Title: Chemotherapy (Paclitaxel and Carboplatin)and Thoracic Radiotherapy With Swallowed Manganese Superoxide Dismutase (MnSOD) Plasmid Liposome Protection in Patients With Locally Advanced Stage III Non-Small Cell Lung Cancer: A Phase I-II Study
Brief Title: MnSOD (Esophageal Protectant) to Prevent Esophagitis During Radiation/Chemotherapy Treatment for Non-Small Cell Lung Cancer (NSCLC)
Acronym: MnSOD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: MnSOD longer available during Phase II
Sponsor: Joel Greenberger (Other)
Responsible Party: Sponsor-Investigator, Joel Greenberger, Professor, Chairman of Radiation Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-054; UPCI 01-054 (Other: University of Pittsburgh Cancer Institute)
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-10

CONDITIONS: Esophageal; Toxicity
Keywords: NSCLC; lung cancer; chemotherapy; radiation therapy; radiation toxicity
MeSH Terms: conditions — Lung Neoplasms; Radiation Injuries | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Radiation + MnSOD PL + Paclitaxel + Carboplatin (Experimental): MnSOD PL (0.3, 3, or 30 mg) + (Paclitaxel + Carboplatin (45mg/m^2)) + Radiation 1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.
  Interventions: Genetic: Manganese Superoxide Dismutase Plasmid Liposome; Drug: carboplatin; Drug: paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Genetic: Manganese Superoxide Dismutase Plasmid Liposome — 15 ml of liquid that contains either 0.3 mg, 3.0 mg or 30.0 mg (depending on which cohort is open when the subject is entered) of MnSOD PL This will be given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  Other Names: MnSOD/PL
Drug: carboplatin — Chemotherapy to stop the growth of tumor cells.
  Other Names: Paraplatin
Drug: paclitaxel — Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
  Other Names: Taxol
Radiation: Radiation Therapy — 1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.

SUMMARY:
This is a Phase I-II study evaluating the feasibility, safety, and efficacy of swallowed MnSOD plasmid/liposome (PL) transgene given as protection against radiation-induced esophagitis during concurrent paclitaxel and carboplatin chemotherapy with thoracic radiation in subjects with locally advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase I-II study evaluating the feasibility, safety, and efficacy of swallowed MnSOD plasmid/liposome (PL) transgene given as protection against radiation-induced esophagitis during concurrent paclitaxel and carboplatin chemotherapy with thoracic radiation in subjects with locally advanced non-small cell lung cancer (NSCLC). Phase I of the study will assess the feasibility and safety of MnSOD PL by dose escalation in 3 cohorts of 3 chemoradiotherapy subjects each (Cohort1 = 0.3 mg/dose, Cohort2 = 3 mg/dose, Cohort3 = 30 mg/dose). The highest dose completed (as determined by toxicity monitoring for 8 weeks from initial treatment) will be the starting dose for Phase II. Phase II will examine the efficacy of MnSOD PL by assessing the incidence of Grade 3 or 4 esophagitis in 27 additional chemoradiotherapy subjects. Incidence of esophageal toxicity, as well as clinical response to the combination of chemoradiotherapy with MnSOD PL are the outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC including squamous cell carcinoma, adenocarcinoma (including bronchoalveolar cell), and large cell anaplastic carcinoma (including giant and clear cell carcinomas) and poorly differentiated non-small cell lung cancer. Totally resected tumors are excluded.
* Subjects must be without evidence of M0.
* Subjects with T1 or T2 disease with N2 or tumor stage 3, lymph node metastasis 1-2 ( stage 1) disease (Stage IIIA) are eligible if they are medically inoperable. Subjects with T4 with any N or any T with N3 disease are eligible. Radiographic evidence of mediastinal lymph nodes >2.0 cm in the largest diameter is sufficient to stage N2 or N3 disease. If the largest mediastinal node is < 2.0 cm in diameter and this is the basis for stage III disease, then at least one of the nodes must be proven positive cytologically or histologically.
* Subjects with tumors adjacent to a vertebral body are eligible as long as all gross disease can be encompassed in the radiation boost field. The boost volume must be limited to < 50% of the ipsilateral lung volume.
* Subjects with a pleural effusion that is a transudate, cytologically negative and non-bloody are eligible if the radiation oncologists feel the tumor can still be encompassed within a reasonable field of radiotherapy. Exudative, bloody, or cytologically malignant effusions are ineligible. If a pleural effusion can be seen on the chest CT but not on chest X-ray and is too small to tap, the subject will be eligible.
* Subjects must be deemed a suitable candidate for protocol treatment by both Radiation Oncology and Medical Oncology
* Subjects must have a Performance Status > 70 (Karnofsky Performance Scale).
* Subjects Weight loss < 10% in 3 months prior to diagnosis.
* Subjects must be male or female > 18 years.
* Subjects must have had no prior systemic chemotherapy, radiation therapy to the thorax, or total surgical resection.
* At least 3 weeks since formal exploratory thoracotomy and the subject has recovered from surgery, or 1 week from diagnostic thoracoscopy.
* Laboratory values must be as follows: (See Section 6.1 of the full protocol for required timing): Granulocytes > 2,000/ml, Platelets > 100,000/ml, Hemoglobin* > 8 mg/dl, Bilirubin < 1.5 x normal, Creatinine clearance > 50 ml/n (24 hour or calculated, forced expiratory volume at one second > 800 cc. Note: *Physician can maintain a subject's hemoglobin with the use of Erythropoetin or transfusions prophylactic use of G-CSF (colony stimulating factor, is not permitted).
* Subjects must have a MRI or CT brain scan within 4 weeks prior to study entry to rule out asymptomatic brain metastases.
* Subjects must be informed of the investigational nature of the study and sign an informed consent form and have no serious medical or psychiatric illnesses that would prevent informed consent.
* No history of serious cardiac disease that is not adequately controlled.
* Female subjects must be non-pregnant and non-lactating. Female subjects of childbearing potential must implement an effective method of contraception during the study. All women of childbearing potential must have a pre-study negative serum or urine pregnancy test within 7 days prior to study entry.

Exclusion Criteria

* Inability to meet any of the above eligibility requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-11-11 (Actual); Primary Completion 2010-02-26 (Actual); Study Completion 2011-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Greenberger, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin: MnSOD PL (0.3 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that containing 0.3 mg of MnSOD PL, given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  Paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
  Carboplatin: Chemotherapy to stop the growth of tumor cells.
- MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin: MnSOD PL (3.0 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that containing 3.0 mg of MnSOD PL, given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  Paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
  Carboplatin: Chemotherapy to stop the growth of tumor cells.
- MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin: MnSOD PL (30.0 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that containing 30.0 mg of MnSOD PL, given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  Paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
  Carboplatin: Chemotherapy to stop the growth of tumor cells.
Period: Overall Study
Arm/Group | MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin | MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin | MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin
Started | 4 | 3 | 11
Completed | 3 | 3 | 11
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients that received at least one dose of MnSOD.
Groups:
- Radiation + MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin: Radiation + MnSOD PL (0.3 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that contains 0.3 mg of MnSOD PL, given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
- Radiation + MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin: Radiation + MnSOD PL (3.0 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that contains 3.0 mg of MnSOD PL, given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
- Radiation + MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin: Radiation + MnSOD PL (30.0 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that contains 30.0 mg of MnSOD PL, given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
- Total: Total of all reporting groups
Arm/Group | Radiation + MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin | Radiation + MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin | Radiation + MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 4 | 3 | 11 | 18
Age, Continuous [Median (Full Range); unit: years] | 62 [50 to 75] | 70 [55 to 75] | 64 [49 to 78] | 65 [49 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 5 | 7
  Male | 3 | 2 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 11 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Determination of Recommended Phase II Dose of MnSOD/Plasmid DNA
Description: The maximally tolerated dose (milligrams) defined as the highest dose with fewer than one-third of patients experiencing a dose-limiting toxicity (DLT) per CTCAE v3.0 due to MnSOD.
  (Three patients treated at each at three tiers of 0.3, 3, and 30mg of MnSOD/plasmid DNA. If no DLTs (grade III/IV toxicity due to MnSOD PL) observed, the dose of MnSOD PL escalated to the next tier. If one DLT observed, the cohort is expanded to six patients. If two of six patients experienced a DLT, dose escalation stops and the next lowest dose declared maximum tolerated dose (MTD). If none of three or one of six patients experience DLT at the 30-mg tier, that dose is defined as the starting dose for the efficacy phase and the MTD would be undefined).
Time Frame: Every 8 weeks, up to 2 years
Population: Patients that received at least one dose of MnSOD.
Measure: Number; unit: milligrams
Groups:
- Radiation + MnSOD PL + Paclitaxel + Carboplatin: Radiation: 1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.
  MnSOD PL (0.3, 3, or 30 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that contains either 0.3 mg, 3.0 mg or 30.0 mg (depending on which cohort is open when the subject is entered) of MnSOD PL This will be given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
Arm/Group | Radiation + MnSOD PL + Paclitaxel + Carboplatin
Number analyzed (Participants) | 18
milligrams | 30

2. Primary Outcome: Radiation-induced Esophageal Toxicity
Description: Number of patients experiencing grade III/IV esophageal toxicity per CTCAE v3.0.
Time Frame: Up to 2 years
Population: Patients treated at 30mg MnSOD (the phase II dose).
Measure: Count of Participants; unit: Participants
Groups:
- Radiation + MnSOD PL + Paclitaxel + Carboplatin: Radiation + MnSOD PL (30 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Radiation: 1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that contains 30.0 mg of MnSOD PL on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
Arm/Group | Radiation + MnSOD PL + Paclitaxel + Carboplatin
Number analyzed (Participants) | 8
Participants | 0

3. Secondary Outcome: Overall (Objective) Response
Description: Clinical Response per Response Evaluation Criteria in Solid Tumors (RECIST). Per RECIST v1.0: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease: Neither sufficient shrinkage (compared to baseline) to qualify for partial or complete response (CR or PR) nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD). Progressive Disease (PD): At least a 20%increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 2 years
Population: Patients that received 30.0 mg MnSOD and evaluable for response.
Measure: Count of Participants; unit: Participants
Groups:
- MnSOD PL + Paclitaxel + Carboplatin: Radiation + MnSOD PL (30 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Radiation: 1.9-2.1 Gy daily 5 times per week (4-6 hr after the first MnSOD PL dose). The total dose planned at 77.0 Gy with a range of 69-84Gy in 34-38 fractions over 7-8 weeks.
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that contains 30.0 mg of MnSOD PL on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
Arm/Group | MnSOD PL + Paclitaxel + Carboplatin
Number analyzed (Participants) | 8
Participants
  Partial Response per RECIST | 3
  Stable Disease per RECIST | 2
  Progressive Disease per RECIST | 2

4. Secondary Outcome: Overall Survival (OS)
Description: The length of time from start of treatment that diagnosed patients remain alive.
Time Frame: Up to 5 years
Population: Patients that received 30.0 mg MnSOD (may or may not have been evaluable for response).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Radiation + MnSOD PL + Paclitaxel + Carboplatin
Number analyzed (Participants) | 8
months | 31 [NA to NA] — CI not reached due to low patient accrual.

5. Secondary Outcome: Time to Disease Progression
Description: The length of time from start of treatment until patients first disease recurrence/progression. Per RECIST v1.0: Progressive Disease (PD): At least a 20%increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 5 years
Population: Patients who received 30.0 mg of MnSOD and were evaluable for response.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Radiation + MnSOD PL + Paclitaxel + Carboplatin
Number analyzed (Participants) | 7
months | 26 [15.3 to NA] — Upper bound of CI not reached due to low patient accrual.

ADVERSE EVENTS:
Time Frame: Adverse Events monitored for up to 2 years; All-Cause Mortality monitored for up to 5 years, defined as a Grade 5 event per CTCAE v3.0
Description: NCI Common Terminology Criteria for Adverse Events CTCAE v 3.0 - Adverse Events: Grade 1 and Grade 2 events per CTCAE v3.0 Serious Adverse Events: Grade 3 and Grade 4 events per CTCAE v3.0
Groups:
- MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin: MnSOD PL (0.3 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that containing 0.3 mg of MnSOD PL This will be given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
- MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin: MnSOD PL (3.0 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that containing 3.0 mg of MnSOD PL This will be given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
- MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin: MnSOD PL (30.0 mg) + (Paclitaxel + Carboplatin (45mg/m^2))
  Manganese Superoxide Dismutase Plasmid Liposome: 15 ml of liquid that containing 30.0 mg of MnSOD PL This will be given on Day 1 and 3 of each week of the experimental treatment for a total of 14 doses.
  carboplatin: Chemotherapy to stop the growth of tumor cells.
  paclitaxel: Chemotherapy to stop the growth of tumor cells. This drug kills tumor cells by inducing multipolar divisions. Cells entering mitosis in the presence of concentrations of paclitaxel equivalent to those in human breast tumors form abnormal spindles that contain additional spindle poles.
Arm/Group | MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin | MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin | MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/3 | 7/11
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin (N=4) | MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin (N=3) | MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin (N=11)
Thrombosis/embolism (Vascular disorders) | 1 | 0 | 0
Cardiovascular/General-Other (Vascular disorders) | 1 | 0 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Gastrointestinal disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Confusion (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 6
Supraventricular and nodal arrhythmia, Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Vasovagal episode (Cardiac disorders) | 0 | 0 | 1
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 0 | 0 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 0 | 2
Hemorrhage, GI, Rectum (Gastrointestinal disorders) | 0 | 0 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Syncope (fainting) (Nervous system disorders) | 0 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MnSOD PL (0.3 mg) + Paclitaxel + Carboplatin (N=4) | MnSOD PL (3.0 mg) + Paclitaxel + Carboplatin (N=3) | MnSOD PL (30.0 mg) + Paclitaxel + Carboplatin (N=11)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0 | 0
Edema (Cardiac disorders) | 1 | 0 | 0
Fatigue (lethargy, malaise, asthenia) (General disorders) | 3 | 0 | 0
Weight loss (General disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia-pharyngeal related to radiation (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 2 | 0 | 0
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 3 | 0 | 0
Infection without neutropenia (Infections and infestations) | 1 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 1 | 0 | 0
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 1 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 8
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 | 0 | 8
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 5
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 | 0 | 8
Platelets (Blood and lymphatic system disorders) | 0 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 1
Supraventricular and nodal arrhythmia, Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Supraventricular and nodal arrhythmia, Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Hypertension (Cardiac disorders) | 0 | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1 | 0
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 0 | 0 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 3 | 8
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 | 0 | 1
Insomnia (General disorders) | 0 | 1 | 1
Sweating (diaphoresis) (General disorders) | 0 | 0 | 1
Weight loss (General disorders) | 0 | 0 | 2
Flushing (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash: dermatitis associated with radiation, Radiation (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 3
Dehydration (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 1 | 6
Esophagitis (Gastrointestinal disorders) | 0 | 2 | 6
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 0 | 1 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 0 | 5
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 | 0 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 | 0 | 3
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 | 0 | 3
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 2
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Glomerular filtration rate (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 9
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 0 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 4
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 | 1 | 0
Neuropathy: sensory (Nervous system disorders) | 0 | 1 | 0
Pain, Chest wall (General disorders) | 0 | 1 | 0
Pain, Chest/thorax NOS (General disorders) | 0 | 1 | 1
Pain, Esophagus (General disorders) | 0 | 0 | 1
Pain, Extremity-limb (General disorders) | 0 | 0 | 2
Pain, Head/headache (General disorders) | 0 | 0 | 2
Pain, Joint (General disorders) | 0 | 1 | 0
Pain, Muscle (General disorders) | 0 | 0 | 2
Pain, Throat/pharynx/larynx (General disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT00618917/Prot_SAP_000.pdf